CLINICAL TRIAL: NCT02598193
Title: An Exploratory Multicenter, Open-Label, Single Arm Study of the Safety and Tolerability of Pirfenidone (Esbriet®) in Combination With Nintedanib (Ofev®) in Patients With Idiopathic Pulmonary Fibrosis
Brief Title: Safety and Tolerability Study of Pirfenidone in Combination With Nintedanib in Participants With Idiopathic Pulmonary Fibrosis (IPF)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA29895; 2015-003280-11 (EudraCT Number)
Record Dates: First submitted 2015-11-04; First posted 2015-11-05 (Estimated); Results first posted 2018-06-13 (Actual); Last update posted 2018-06-13 (Actual); Status verified 2018-05

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — nintedanib; pirfenidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pirfenidone+Nintedanib (Experimental): Participants with IPF will receive pirfenidone at 1602-2403 milligrams per day (mg/day) dose and nintedanib at the 200-300 mg/day dose up to 24 weeks.
  Interventions: Drug: Nintedanib; Drug: Pirfenidone

INTERVENTIONS:
Drug: Nintedanib — Participants with IPF will receive nintedanib at the 200-300 mg/day dose up to 24 weeks.
  Other Names: Ofev
Drug: Pirfenidone — Participants with IPF will receive pirfenidone at 1602-2403 mg/day dose up to 24 weeks.
  Other Names: Esbriet

SUMMARY:
This clinical study will evaluate the safety and tolerability of combination treatment of nintedanib and pirfenidone in participants with IPF. Eligible participants must have received pirfenidone for at least 16 weeks on a stable dose. Nintedanib will be added on Day 1 of the study as a combination treatment for IPF for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are on pirfenidone for at least 16 weeks and on a stable dose (defined as 1602-2403 mg/day) for at least 28 days at the start of Screening; the dose must be expected to remain in that range throughout the study
* Documented diagnosis of IPF, per the Investigator per using the criteria of the 2011 American Thoracic Society / European Respiratory Society / Japanese Respiratory Society / Latin American Thoracic Association guidelines
* Participants with percent predicted forced vital capacity (FVC) more than or equal to (>=) 50 percent (%) and percent predicted carbon monoxide diffusing capacity (DLco) >=30% at Screening
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use two adequate methods of contraception, including at least one method with a failure rate of less than (<) 1% per year, during the treatment period and for at least 3 months after the final Follow-up Visit
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures and agreement to refrain from donating sperm during the treatment period and for at least 4 months after the final Follow-up Visit

Exclusion Criteria:

* Participants with clinical evidence of active infection
* Participant with any new or ongoing moderate or severe adverse reaction considered by the Investigator to be related to pirfenidone, or an pirfenidone treatment interruption in the 28 days before the start of Screening
* Any condition that is likely to result in death in the 12 months after the start of Screening
* Lung transplantation anticipated or any planned significant surgical intervention
* Known hypersensitivity to the active substance or any excipient of either pirfenidone or nintedanib
* Mild (Child Pugh A), moderate (Child Pugh B), or severe (Child Pugh C) hepatic and/or severe renal impairment
* History of gastrointestinal (GI) tract perforation, unstable or deteriorating cardiac or pulmonary disease (other than IPF), long QT syndrome, alcohol or substance abuse in the 2 years before the start of screening, use of any tobacco product in the 12 weeks before the start of screening
* Bleeding risk
* Use of Cytochrome P450 (CYP) 1A2 (CYP1A2) inhibitors (for example, fluvoxamine, enoxacin) and/or use of inhibitors of P-glycoprotein (for example, ketoconazole, erythromycin) or CYP3A4 (for example, ketoconazole, erythromycin) or their inducers (for example, rifampicin, carbamazepine, phenytoin, St John's wort) in the 28 days before the start of Screening
* Pregnancy or lactation
* Hypersensitivity to peanuts and/or soy
* Use of pirfenidone and/or nintedanib in a clinical study protocol in the 28 days before the start of screening

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2016-01-14 (Actual); Primary Completion 2017-05-16 (Actual); Study Completion 2017-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (38):
- United States (16):
  - David Geffen School of Medicine at UCLA;Division of Pulmonary & Critical Care/ Department of Medic, Los Angeles, California
  - Stanford University School of Medicine ; Pulmonary/Critical Care Medicine, Stanford, California
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Cardio-Pulmonary Associates of St. Luke's Hospital, Chesterfield, Missouri
  - Creighton University, Omaha, Nebraska
  - Atlantic Respiratory Institute, Summit, New Jersey
  - Mount Sinai School of Medicine, New York, New York
  - Columbia University Medical Center, New York, New York
  - Pulmonix LLC, Greensboro, North Carolina
  - UC Health Clinical Trials Office, Cincinnati, Ohio
  - John A. Butler, M.D. - Oregon Pulmonary Associates, Portland, Oregon
  - Medical University of South Carolina (MUSC); MUSC Pulmonary, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Inova Health Care Services; Advanced Lung Disease Transplant Program, Falls Church, Virginia
- Canada (2):
  - South Health Campus/Alberta Health Services/ University of Calgary, Calgary, Alberta
  - University Health Network, Toronto, Ontario
- Gentofte Hospital, Lungemedicinsk Afdeling, Hellerup, Denmark
- France (3):
  - Hopital Avicenne; Pneumologie, Bobigny
  - Hopital Louis Pradel; Pneumologie, Bron
  - Hopital de Pontchaillou; Service de Pneumologie, Rennes
- Germany (3):
  - Fachkrankenhaus Coswig GmbH Zentrum f.Pneumologie Beatmungsmedizin Thorax-u.Gefäßchirurgie, Coswig
  - Ruhrlandklinik Lungenzentrum der UNI Essen Abt.Pneumologie-Allergologie, Essen
  - Klinikum Fulda gAG; Universitätsmedizin Marburg, Campus Fulda, Fulda
- Italy (4):
  - ASST DI MONZA; U O Clinica Pneumologica, Monza, Lombardy
  - A.O. Universitaria San Luigi Gonzaga di Orbassano; Malattie Apparato Respiratorio (MAR2), Orbassano, Piedmont
  - Azienda Ospedaliero Universitaria Pisana; U.O. Pneumologia, Pisa, Tuscany
  - A.O. Univ. Senese Policlinico S. Maria alle Scotte; UOC Malattie Resepiratorie e Trapianto Polmonare, Siena, Tuscany
- Netherlands (2):
  - Antonius Ziekenhuis; Dept of Lung Diseases, Nieuwegein
  - Erasmus MC; Afdeling Longziekten, Rotterdam
- Spain (7):
  - Hospital Universitari de Bellvitge ; Servicio de Neumologia, L'Hospitalet de Llobregat, Barcelona
  - Hospital del Henares; Medicina Interna. Unidad de Neumología, Coslada (Madrid), Madrid
  - Hospital Universitario de Canarias; Servicio de Neumologia, San Cristóbal de La Laguna, Tenerife
  - Complejo Asistencial Universitario de Leon; Pneumology, León
  - Hospital Universitario La Princesa; Servicio de Neumologia, Madrid
  - Hospital Universitario Virgen del Rocio; Servicio de Neumologia, Seville
  - Hospital General Universitario De Valencia; Servicio de Neumologia, Valencia

REFERENCES:
- [Derived] Flaherty KR, Fell CD, Huggins JT, Nunes H, Sussman R, Valenzuela C, Petzinger U, Stauffer JL, Gilberg F, Bengus M, Wijsenbeek M. Safety of nintedanib added to pirfenidone treatment for idiopathic pulmonary fibrosis. Eur Respir J. 2018 Aug 2;52(2):1800230. doi: 10.1183/13993003.00230-2018. Print 2018 Aug. PMID 29946005

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with idiopathic pulmonary fibrosis were recruited for this study.
Pre-assignment Details: At the start of screening, participants were on pirfenidone for at least 16 weeks and on a stable dose (1602-2403 mg/d) for at least 28 days. A total of 109 participants were screened, 20 participants were screen failures and 89 were enrolled at 36 study centers in 8 countries.
Groups:
- Pirfenidone+Nintedanib: Participants with idiopathic pulmonary fibrosis (IPF) received pirfenidone at 1602-2403 milligrams per day (mg/day) dose and nintedanib at the 200-300 mg/day dose up to 24 weeks.
Period: Overall Study
Arm/Group | Pirfenidone+Nintedanib
Started | 89
Completed | 73
Not Completed | 16
Not completed — Adverse Event | 13
Not completed — Withdrawal by Subject | 1
Not completed — Listed in active lung transplant list | 1
Not completed — Does not want to take Nintedanib | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who had received at least one dose of investigational medicinal product on or after Day 1.
Arm/Group | Pirfenidone+Nintedanib
Number analyzed (Participants) | 89
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.2 (6.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 74
  Unknown or Not Reported | 6
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 84
  Black or African American | 3
  Asian | 1
  Asian/White | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Complete 24 Weeks of Combination Treatment on Pirfenidone at a Dose of 1602-2403 mg/Day and Nintedanib at a Dose of 200-300 mg/Day
Time Frame: Week 24
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pirfenidone+Nintedanib
Number analyzed (Participants) | 89
Percentage of Participants | 77.5 [67.4 to 85.7]

2. Secondary Outcome: Percentage of Participants With Adverse Events and Serious Adverse Events
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Baseline up to Week 28
Population: as for baseline characteristics
Measure: Number; unit: Percentage of Participants
Arm/Group | Pirfenidone+Nintedanib
Number analyzed (Participants) | 89
Percentage of Participants
  Adverse Event | 98.9
  Serious Adverse Event | 18.0

3. Secondary Outcome: Percentage of Participants Who Discontinue Pirfenidone, Nintedanib, or Both Study Treatments Because of Adverse Events Before the Week 24 Visit
Time Frame: Baseline up to Week 24
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of Praticipants
Arm/Group | Pirfenidone+Nintedanib
Number analyzed (Participants) | 13
Percentage of Praticipants | 14.6 [8.0 to 23.7]

4. Secondary Outcome: Total Number of Participant Days of Combination Treatment With Pirfenidone and Nintedanib
Time Frame: Baseline up to Week 24
Population: as for baseline characteristics
Measure: Number; unit: Participant Days
Arm/Group | Pirfenidone+Nintedanib
Number analyzed (Participants) | 89
Participant Days | 13330

5. Secondary Outcome: Total Number of Days From the Initiation of Combination Treatment to Discontinuation of Pirfenidone, Nintedanib, or Both Study Treatments
Time Frame: Baseline up to Week 24
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Number of Days
Arm/Group | Pirfenidone+Nintedanib
Number analyzed (Participants) | 89
Number of Days | 149.8 (43.93)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 28
Description: Safety population included all participants who had received at least one dose of investigational medicinal product on or after Day 1.
Arm/Group | Pirfenidone+Nintedanib
All-Cause Mortality (participants affected / at risk) | 0/89
Serious Adverse Events (participants affected / at risk) | 16/89
Other Adverse Events (participants affected / at risk) | 83/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pirfenidone+Nintedanib (N=89)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cholecystitis infective (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Tracheobronchitis (Infections and infestations) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pirfenidone+Nintedanib (N=89)
Diarrhoea (Gastrointestinal disorders) | 52 (184)
Nausea (Gastrointestinal disorders) | 44 (70)
Vomiting (Gastrointestinal disorders) | 29 (57)
Dyspepsia (Gastrointestinal disorders) | 8 (8)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 (7)
Abdominal pain upper (Gastrointestinal disorders) | 6 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 20 (22)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Headache (Nervous system disorders) | 13 (22)
Dizziness (Nervous system disorders) | 9 (9)
Fatigue (General disorders) | 14 (16)
Non-cardiac chest pain (General disorders) | 5 (6)
Viral upper respiratory tract infection (Infections and infestations) | 9 (13)
Upper respiratory tract infection (Infections and infestations) | 8 (9)
Decreased appetite (Metabolism and nutrition disorders) | 14 (14)
Weight decreased (Investigations) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-05-17): https://cdn.clinicaltrials.gov/large-docs/93/NCT02598193/SAP_000.pdf
  • Study Protocol (2016-06-21): https://cdn.clinicaltrials.gov/large-docs/93/NCT02598193/Prot_001.pdf